CLINICAL TRIAL: NCT05930938
Title: A Double-blind, Randomized, Phase III Study of Radiotherapy Combined With cetuXimab + Xevinapant Compared to Radiotherapy Combined With Cetuximab (Standard of Care) + Placebo in Patients With LA SCCHN, Unfit for High-dose Cisplatin
Brief Title: Study Comparing RT With Cetuximab + Xevinapant to RT With Cetuximab-placebo in Patients With Head and Neck Cancer
Acronym: XXL_2022-01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: toxicity
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-502584-38-00
Record Dates: First submitted 2023-06-23; First posted 2023-07-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: Participants who meet the study criteria will be randomly assigned in a 1:1 ratio using minimization to Arm A or arm B
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-RT-cetuximab (Placebo Comparator): 3 cycles of placebo (matching oral solution from Day 1 to 14, per 3-week cycle) + IMRT (69.96 Gy in 33 fractions, 2.12 Gy/fraction) + cetuximab (loading dose of 400 mg/m² IV on Day -7, followed by weekly dose of 250 mg/m² IV until the end of the RT), followed
  Interventions: Drug: Placebo; Drug: cetuximab; Radiation: IMRT
- Xevinapant-RT-cetuximab (Experimental): 3 cycles of xevinapant (oral solution 200 mg/day from Day 1 to 14, per 3-week cycle) + IMRT (69.96 Gy in 33 fractions, 2.12 Gy/fraction) + cetuximab (loading dose of 400 mg/m² IV on Day -7, followed by weekly dose of 250 mg/m² IV until the end of the RT), followed by 3 cycles of monotherapy of xevinapant (200 mg/day from Day 1 to 14, per 3-week cycle)
  Interventions: Drug: Xevinapant; Drug: cetuximab; Radiation: IMRT

INTERVENTIONS:
Drug: Xevinapant — Xevinapant is a multi-IAP antagonist that blocks the activity of several IAPs including X-linked IAP (XIAP), cellular inhibitor of apoptosis proteins (cIAP) 1, cIAP2 and ML-IAP
  Arms: Xevinapant-RT-cetuximab
Drug: Placebo — Xevinapant without active substance
  Arms: Placebo-RT-cetuximab
Drug: cetuximab — cetuximab
Radiation: IMRT — IMRT (69.96 Gy in 33 fractions, 2.12 Gy/fraction)

SUMMARY:
Xevinapant is an antagonist of inhibitor of apoptosis proteins (IAPs) that has been shown both chemo-, radiosensitizing, and immunomodulatory activities in nonclinical in vitro and in vivo squamous cell carcinoma of the head and neck (SCCHN) models. In previously untreated patients with non-resected locally advanced SCCHN, the addition of xevinapant recently showed a significant improvement of progression-free survival (PFS), overall survival (OS) and loco-regional control at 3 years after completing treatment. Thus, the purpose of this Phase III study is to demonstrate the superior efficacy to the xevinapant when it is administered in combination with radiotherapy (RT)+cetuximab compared to radiotherapy+cetuximab (SoC) + placebo in previously untreated participants with LA-SCCHN, ineligible for high-dose cisplatin defined as ≥ 200 mg/m² (projective total cumulative dose) throughout the course of the radiotherapy.

DETAILED DESCRIPTION:
CT-RT and especially cisplatin-RT is a well-established and the most commonly used SoC for patients with LA SCCHN15. However, a large proportion of patients with LA SCCHN are not suitable for high dose platin based CT-RT for several reasons (age, medical/general conditions and or comorbidities…).

Based on recent GORTEC study, the proportion of patients unfit for receiving high-dose of cisplatin was 43% among 707 patients randomized19. In the corresponding cohort of the REACH study, the characteristics of the population (same population to be included in the XXL study) were fragile patients, unfit for high-dose cisplatin, with heavy alcohol and tobacco consumption, numerous comorbidities and a median age 67 years. In this population, there was a trend in the triplet combination of cetuximab-avelumab-RT towards improving PFS, but the triplet was also associated with increased death without previous cancer progression in the first 6 months after RT. In the control arm, the doublet of cetuximab-RT regimen was better tolerated with no excess of death. Same good tolerance was also observed with doublet treatments in both arms of the PembroRad trial (NCT02707588).

The addition of xevinapant to cetuximab is combining two complementary radiosensitizing effects that could ultimately improve the tumor control when compared to cetuximab alone. However, it is

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female ≥ 18 years (or based on the country legal age limit for adults on day of signing the Informed Consent Form, ICF) and < 80 years
2. ECOG PS 0-1
3. Histologically confirmed diagnosis in previously untreated LA-SCCHN participant (Stage III, IVA or IVB according to the American Joint Committee on Cancer-TNM Staging System, 8th Ed.) of at least one of the following sites: oral cavity, hypopharynx and larynx. OPC participants are also eligible but their primary tumor must be:

   * HPV-negative (Stage III, IVA or IVB according to the American Joint Committee on Cancer/TNM Staging System, 8th Ed.) or
   * HPV-positive and smokers > 20 PY and must have according to the American Joint Committee on Cancer/TNM Staging System, 8th Ed:

     * T3 N1-3
     * T4 and any N Note: HPV status is determined by p16 expression using IHC (pathological report should be available).

   Note: Patient with primary tumor of unknown primary site are not eligible.
4. Able to swallow liquids or have an adequately functioning feeding tube, gastrostomy or jejunostomy placed.
5. Patients must be ineligible to receive high-dose cisplatin defined as ≥ 200 mg/m² (projected total cumulative dose throughout the course of the RT). Ineligibility is defined as at least one of the following criteria:

   * eGFR < 60 mL/min /1.73 m² (using the CKD-EPI creatinine formula)
   * History of hearing loss, defined as either:

     i. Existing need of a hearing aid and/or ii. Clinically relevant hearing loss by clinical assessment including tinnitus ≥ Grade 2. Note: In case of doubt, an audiogram should be requested to guide the Investigator
   * Peripheral neuropathy ≥ Grade 2
   * Cardiac function not compatible with hyperhydration
   * If > 70 years, unfit according to G8 questionnaire (Score ≤ 14)
6. Adequate hematologic, renal and hepatic function as indicated by (using CTCAE v5.0):

   * Absolute neutrophil count ≥ 1500 /mm3
   * Platelets ≥ 100 000 /mm3
   * Hemoglobin ≥ 9.0 g/dL (blood transfusions during Screening are not permitted)
   * White blood cells ≥ 3 000/mm3
   * AST and ALT ≤ 3 × ULN
   * eGFR ≥ 30 mL/min /1.73 m² (using the CKD-EPI creatinine formula)
   * Total bilirubin ≤ 1.5 × ULN (up to 2.0 × ULN is allowed if the direct bilirubin level is normal, and the elevation is limited to indirect bilirubin)
7. The Investigator confirms that the participant agrees to use appropriate contraception and barriers methods, if applicable. The contraception, barrier, and pregnancy testing requirements are below:

   -A female participant: i. Is not a WOCBP, no need serum pregnancy test or contraceptive method ii. If WOCBP, she must agree to use a highly effective contraceptive method (i.e., with a failure rate of < 1% per year), preferably with low user dependency, as described in section 3.3 from Inform Consent Form (ICF) to at least 6 months after the last dose of cetuximab or 3 months after the last dose of xevinapant/placebo, whichever is the latest. WOCBP must not agree to donate eggs (ova, oocytes) for reproduction during this period. Female participants using hormonal contraception must also use a barrier contraception method (preferably male condom) due to potential risk of CYP3A4 induction by xevinapant which may reduce hormonal contraception efficacy.

   Note: The investigator evaluates the effectiveness of the contraceptive method in relationship to the date of randomization. The Investigator reviews the medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a female with an early undetected pregnancy.

   -A male participant must agree to the following from ICF signature to at least 6 months after the last dose of cetuximab or 3 months after the last dose of xevinapant/placebo, whichever is the latest: i. To refrain from donating fresh unwashed semen. If not done previously, cryopreservation of sperm prior to receiving study treatments is advised to male patients with a desire to have children.

   ii. Non-sterilized males who are sexually active with a female partner of childbearing potential must agree to use condom and spermicide. Because male condom and spermicide is not a highly effective contraception method, it is required that female partners of a male study participant use a highly effective contraceptive method (with a failure rate of < 1% per year, as described in section 3.3).
8. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the inform consent form and this protocol.

Exclusion Criteria:

1. Any condition, including any uncontrolled disease state other than SCCHN that in the Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation.
2. Metastatic disease (according to AJCC/TNM, 8th ed.).
3. Primary tumor of nasopharyngeal, paranasal sinuses, salivary, thyroid or parathyroid gland, skin or unknown primary site.
4. Known history of infection with human immunodeficiency virus (HIV). If unknown history of HIV, an HIV screening test is to be performed and participants with positive serology for HIV-1/2 must be excluded.
5. Known chronically active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. If unknown status, HBV and HCV tests (see section 6.1.2) are to be performed and participants with positive serology must be excluded:

   1. HBV screening tests: both HBV Ag and Anti-HepB core IgG.
   2. HCV screening tests: both HCV-antibody and positive viral load HCV-RNA by PCR. Note: Positive serology is defined as the presence of hepatitis B core antibody [anti-HBc] and/or presence of HBsAg and/or the presence of HCV antibody and/or positive for HCV RNA by PCR.
6. Other infections (viral [including COVID-19] and/or mycotic) requiring systemic treatment.
7. Ongoing uncontrolled infection requiring intravenous antibiotic therapy within 7 days prior to randomization.
8. Known gastrointestinal disorder with clinically established malabsorption syndrome and major gastrointestinal surgery that may limit oral absorption.
9. Documented weight loss of > 10% during the last 4 weeks prior to randomization (unless adequate measures are undertaken for nutritional support), OR plasmatic albumin < 3.0 g/dL. No albumin transfusions are allowed within 2 weeks before randomization.
10. Active gastrointestinal bleeding, or any other uncontrolled bleeding requiring more than 2 red blood cell transfusions or 4 units of packed red blood cells within 4 weeks prior to randomization.
11. Active uncontrolled inflammatory disease (including rheumatoid arthritis, systemic lupus erythematosus, Sjögren syndrome, severe extensive psoriasis, and other autoimmune diseases) requiring ongoing treatment with anti-TNF medication.
12. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

    1. Ongoing or history of uncontrolled or symptomatic ischemic myocardiopathy within 6 months prior to randomization.
    2. Known left ventricular ejection fraction < 50%, left ventricular hypertrophy, ventricular arrhythmias, bradycardia (heart rate < 50 bpm).
    3. History of myocardial infarction, or severe/unstable angina, within 6 months prior to randomization.
    4. New York Heart Association Class > 2 congestive heart failure.
    5. Congenital long QT syndrome.
    6. Family history of long QT syndrome.
    7. Symptomatic pulmonary embolism within 6 months prior to randomization.
    8. Ongoing or known history of transient ischemic attacks or stroke within 6 months prior to randomization.
    9. QTc using Fridericia's formula (QTcF) interval > 450 ms for males and > 470 ms for females.
13. Hypertension uncontrolled by medication (i.e. systolic blood pressure > 150 mmHg and diastolic blood pressure > 90 mmHg).
14. Symptomatic pulmonary disease requiring continuous or intermittent oxygen supply.
15. History of another malignancy within the last 3 years prior to randomization, with the exception of completely resected non-melanoma cell skin cancer outside the head and neck area or completely resected stage I breast cancer, or completely resected in-situ non-muscular invasive bladder, cervix and/or uterine carcinomas.
16. Non compensated or symptomatic liver cirrhosis (Child-Pugh score: B or C).
17. Current alcohol and/or drug abuse that puts at risk the compliance to the study procedures in the opinion of the Investigator.
18. Prior definitive or adjuvant RT and/or radical surgery to the head and neck region which may jeopardize the primary tumor irradiation plan in the opinion of the Investigator, or any other prior systemic treatment for SCCHN, including investigational agents.
19. Use within 14 days prior to randomization or requirement for ongoing treatment with any drug(s) on the prohibited medication list (see section 4.5.2 of the protocol).
20. Treatment with an investigational agent or use of an investigational device within 4 weeks of the first dose of study treatment.
21. Any concomitant medication known to prolong the QT interval that cannot be discontinued or replaced by safe alternative medication within 7 days prior to start of treatment.
22. Concurrent use of anticancer therapy.
23. Previous treatment with or hypersensitivity to cetuximab or other eGFR targeting agents or to monoclonal antibodies.
24. Major surgical intervention within 4 weeks prior to the first dose of study intervention. Biopsy(s) to establish the diagnosis for SCCHN is permitted.
25. Prior organ transplantation, including allogeneic stem cell transplantation.
26. Participation in any clinical interventional study within 28 days prior to screening or during participation in this study.
27. Known allergy to xevinapant, cetuximab, monoclonal antibodies, or any excipient known to be present in xevinapant formulation.
28. Pregnant or nursing (lactating) women.
29. Patient under guardianship, curatorship or deprived of liberty

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | through study completion, an average of 1 year"
  PFS as assessed by independent review committee (IRC) defined as the time from randomization to the first occurrence of any of the following events: death from any cause, disease progression (PD), primary treatment failure before achieving a complete response (CR) or any radiological or clinical relapse after achieving a CR.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche Compté, Montbéliard, France